CLINICAL TRIAL: NCT02341872
Title: Compare the Efficacy of the Remineralization Agents on the White Enamel Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ecem Ergin, Dt., Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: thesis
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-05

CONDITIONS: White Spot Lesions
Keywords: White spot lesions; remineralization; QLF; antibacterial
MeSH Terms: interventions — Fluorides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): The investigators won't do any application , the oral hygiene konwledge will be given only.
- Fluoride + Calcium varnish (Active Comparator): The investigators will do fluoride+ calcium varnish( Clinpro White Varnish) application on white spot lesions.
  Interventions: Other: Clinpro White Varnish (fluoride + calcium varnish)
- Polipeptide solution (Experimental): The investigators will do polipeptide ( Curodont Repair) solution application on white spot lesions.
  Interventions: Other: Curodont Repair
- Fluoride + calcium + polipeptide (Experimental): The investigators will do polipeptide ( Curodont Repair) solution and fluoride + calcium varnish (Clinpro White Varnish) application on white spot lesions.
  Interventions: Other: Clinpro White Varnish (fluoride + calcium varnish); Other: Curodont Repair

INTERVENTIONS:
Other: Clinpro White Varnish (fluoride + calcium varnish) — Clinpro White Varnish will be applied to the teeth with brush.
  Arms: Fluoride + Calcium varnish; Fluoride + calcium + polipeptide
Other: Curodont Repair — Curodont Repair solution be applied to the teeth in the form of drops
  Arms: Fluoride + calcium + polipeptide; Polipeptide solution

SUMMARY:
The purpose of this study is to determine whether Fluoride varnish + calcium (Clinpro White Varnish) and polipeptide solution (Curodont Repair) are effective in the treatment of remineralization therapy. The investigators will diagnose their alone or in combination effects on white spot lesions. Aesthetics (tooth-colored), remineralization, microbiological effects will be evaluated separately. Spectrophotometer (Vita Easy Shade) , Quantitative Light Fluorescence (QLF), Diagnodent(Cavo Diagnodent) and culture methods in microbiology laboratories are used for aesthetic, remineralization and microbiological assessments. The measurements will be made baseline, 6 weeks, 3 months and 6 months later after the applications and recorded.

DETAILED DESCRIPTION:
The aim of this study is that evaluate the remineralizing and antibacterial effects of the different remineralization agents. Initiative caries lesions named as white spot lesions and these lesions are localized at enamel. Demineralization is occured but cavitations aren't seen at this stage. It is important to control at this stage with remineralization agents because of the minimally invasive approach.

Fluoride varnish or polipeptide containing agents alone or combination using effects on remineralization, esthetic and bacterial counts will be evaluated with Quantitive Light Fluorescence , Diagnodent (Cavo-Diagnodent), Spectrophotometer (Vita Easy Shade) devices and microbiological assessment at laboratory.

The investigators will choose and include in our study that who come to the Ege University Faculty of Dentistry pediatric department, between 10-18 years olds, healthy and have one or more white spot lesions on her/his permanent teeth.

32 volunteer who have inclusion criteria will be put into pratice. 32 volunteer divided into 4 groups for different applications. We will tell each volunteer that they must brush their teeth twice a day with fluoride dentifrice ( the investigators will give them 1400 ppm fluoride containing fluoride dentifrice)

1. Group: Control group ( The investigators won't do any application , the oral hygiene konwledge will be given only.)
2. Group: Fluoride + Calcium (TCP) (The investigators will do fluoride+ calcium varnish( Clinpro white varnish) application on white spot lesions)
3. Group: Polipeptide solution (The investigators will do polipeptide ( Curodont repair) solution application on white spot lesions)
4. Group: [Fluoride + calcium varnish] + polipeptide solution combination ( The investigators will do polipeptide ( Curodont repair) solution and fluoride + calcium varnish (Clinpro white varnish) application on white spot lesions) First day,the investigators will collect stimulated saliva from each volunteer before any application. Saliva samples will transport to the microbiology laboratory. After any application 6 weeks, 3 months and 6 months later we will collect stimulated saliva again for microbiological assessment.

Nyvad Caries Diagnostic Criteria , ICDAS indexes will be used to make the follow-up of lesions at baseline and 6 months after the application. Plaque index (Silness & Löe , 1964) and bleeding index (Ainamo&Bay ,1976) will be used to assess oral hygiene every visit.

The investigators will use QLF,Diagnodent devices will be used at beginning for evaluate the demineralization level and after applications 6 weeks, 3 months and 6 months later used for evaluate the remineralization level. In addition for determine about esthetic results the investigators will use spectrophotometer (Vita Easy Shade) device at beginning, 6 weeks, 3 months and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* between 10-18 years olds
* healthy
* have one or more white spot lesions on her/his permanent teeth

Exclusion Criteria:

* have any health problem
* unsuitable age
* don't give approval for this study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2013-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
QLF ( ∆F, ∆Q, lesion area) | Change baseline enamel fluorescence level at 6 weeks, 3 and 6 months.
  remineralization level assesment

SECONDARY OUTCOMES:
Salivary Streptococcus mutans and lactobacilli counts | baseline, after 6 weeks, 3 months and 6 months of the application
  Microbiological assesment
Spectrophotometer ( L, a, b) | baseline, after 6 weeks, 3 months and 6 months of the application
  esthetic assesment
Diagnodent | baseline
  remineralization level assesment
Nyvad Caries Diagnostic Criteria index and ICDAS index | baseline
  Evaluation of the state of the lesion

CONTACTS AND LOCATIONS:
Overall Officials: Ecem Ergin, Principal Investigator — Ege University; Ece Eden, Study Director — Ege University; Mustafa Ateş, Study Chair — Ege University
Locations (1):
- Ege University School of Dentistry Department of Pedodontics, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lelli M, Putignano A, Marchetti M, Foltran I, Mangani F, Procaccini M, Roveri N, Orsini G. Remineralization and repair of enamel surface by biomimetic Zn-carbonate hydroxyapatite containing toothpaste: a comparative in vivo study. Front Physiol. 2014 Sep 5;5:333. doi: 10.3389/fphys.2014.00333. eCollection 2014. PMID 25249980
- [Background] Kirkham J, Firth A, Vernals D, Boden N, Robinson C, Shore RC, Brookes SJ, Aggeli A. Self-assembling peptide scaffolds promote enamel remineralization. J Dent Res. 2007 May;86(5):426-30. doi: 10.1177/154405910708600507. PMID 17452562
- [Background] Beerens MW, Boekitwetan F, van der Veen MH, ten Cate JM. White spot lesions after orthodontic treatment assessed by clinical photographs and by quantitative light-induced fluorescence imaging; a retrospective study. Acta Odontol Scand. 2015 Aug;73(6):441-6. doi: 10.3109/00016357.2014.980846. Epub 2014 Nov 25. PMID 25423022
- [Background] Oliveira GM, Ritter AV, Heymann HO, Swift E Jr, Donovan T, Brock G, Wright T. Remineralization effect of CPP-ACP and fluoride for white spot lesions in vitro. J Dent. 2014 Dec;42(12):1592-602. doi: 10.1016/j.jdent.2014.09.004. Epub 2014 Sep 23. PMID 25260438
- [Background] Mehta R, Nandlal B, Prashanth S. Comparative evaluation of remineralization potential of casein phosphopeptide-amorphous calcium phosphate and casein phosphopeptide-amorphous calcium phosphate fluoride on artificial enamel white spot lesion: an in vitro light fluorescence study. Indian J Dent Res. 2013 Nov-Dec;24(6):681-9. doi: 10.4103/0970-9290.127610. PMID 24552927
- [Background] Gomez J, Pretty IA, Santarpia RP 3rd, Cantore B, Rege A, Petrou I, Ellwood RP. Quantitative light-induced fluorescence to measure enamel remineralization in vitro. Caries Res. 2014;48(3):223-7. doi: 10.1159/000354655. Epub 2014 Jan 29. PMID 24481051